CLINICAL TRIAL: NCT02935569
Title: Feasibility Clinical Study of Compression Headband Use to Prevent Hair Loss During Whole Brain Radiotherapy
Brief Title: Compression Headband Use to Prevent Hair Loss During Whole Brain Radiotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results with 4 subjects suggest a redesign of Compression system is required.
Sponsor: Michael Milano, MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Michael Milano, MD,PhD, Assoc Professor, Radiation Oncology, University of Rochester
Organization: University of Rochester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCP12009
Record Dates: First submitted 2012-10-12; First posted 2016-10-17 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Alopecia
Keywords: Alopecia; Radiotherapy
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compression Headband (Experimental): a compression headband, placed only at the time of irradiation
  Interventions: Device: Compression HeadBand

INTERVENTIONS:
Device: Compression HeadBand — * commercially available office rubber bands (Alliance® Sterling Rubber Bands, Size 105) OR commercially available medical non-latex bands (Allegience® 1" x 18" x .025") with Velcro adhesion
  * Plastics disks, hollow (3.5 cm diameter, by 1 cm height)
  Two bands will be placed just behind the ears laterally, and over the occipital protuberance posteriorly. The plastic inserts will be placed in the temporal fossae bilaterally, under the band to provide adequate tension on the temporal artery.

SUMMARY:
This study hypothesizes that in patients undergoing whole brain radiotherapy, a compression headband will decrease the percentage of patients with significant hair loss following radiation.

DETAILED DESCRIPTION:
This is a pilot feasibility study. The primary objective of this study is to seek preliminary information to answer the following question:

1. Does a compression headband, placed only at the time of irradiation, reduce the incidence of significant hair loss after whole brain radiation, as compared to historical controls?

   This study will also seek to answer these secondary questions:
2. Is a temporary compression headband well tolerated in patients undergoing whole brain radiation?
3. If a portion of patients do have significant hair loss after radiation in spite of compression banding, what is the timing of hair regrowth?
4. In normal volunteers, does a compression headband cause acute hypoxia in the scalp, as measured by a transcutaneous oxygen pressure monitor, and, if so, to what degree?

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old.
* Undergoing whole brain radiation therapy, using lateral opposed fields
* Total planned radiation prescription dose between 30 Gy and 37.5 Gy in 10 to 15 treatments.

Exclusion Criteria:

* Current complete or near-complete alopecia (natural or chemotherapy-induced)
* Concurrent or sequential chemotherapy with an agent known to commonly cause alopecia (Adriamycin, Cytoxan, Ifosfamide, Taxol (greater than 50 mg/m2), or Vincristine).
* Previous Radiation to the Scalp
* Any active dermatologic disease affecting the scalp, or temporal arteritis
* History of severe headaches.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in Hair loss defined as grade 1 (thinning or patchy) or grade 2 (complete) alopecia (hair loss), as per Common Toxicity Criteria for Adverse Effects (CTCAE) version 3 | baseline to 6 weeks
  The primary outcome of this study will be the presence of "significant hair loss" by 6 weeks after the completion of whole brain radiation. This will be defined as grade 1 (thinning or patchy) or grade 2 (complete) alopecia (hair loss), as per Common Toxicity Criteria for Adverse Effects (CTCAE) version 3.
  The amount of hair loss will be evaluated at the following time points.
  * Before whole brain radiation
  * six weeks following radiation

SECONDARY OUTCOMES:
Temporary compression headband side effects (Nausea, Headache, Redness, Tingling) in patients undergoing whole brain radiation | 6 weeks
  Does a temporary compression headband cause side effects in patients undergoing whole brain ? Nausea? Headache? Redness? Tingling?
Timing of hair regrowth | one year
  If a portion of patients do have significant hair loss after radiation in spite of compression banding, what is the timing of hair regrowth?
Acute hypoxia in the scalp of normal volunteers caused by compression headband (if present, to what degree?) as measured by a transcutaneous oxygen pressure monitor | 1 hour
  In normal volunteers, does a compression headband cause acute hypoxia in the scalp, as measured by a transcutaneous oxygen pressure monitor, and, if so, to what degree?

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milano, MD, PhD, Principal Investigator — University of Rochester
Locations (1):
- Dept. of Radiation Oncology, University of Rochester, Med Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers can contact the PI to obtain IPD with collaboration.